CLINICAL TRIAL: NCT00884949
Title: A Phase 1/2, Multicenter, Open-label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Efficacy of BMN 110 in Subjects With Mucopolysaccharidosis IVA (Morquio Syndrome)
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of BMN 110 in Subjects With Mucopolysaccharidosis IVA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR-002
Record Dates: First submitted 2009-04-10; First posted 2009-04-21 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: MPS IV A
Keywords: Mucopolysaccharidosis IV type A; MPS IV Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases | interventions — GALNS protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMN 110 (Experimental): Within-patient Dose-Escalation
  Interventions: Drug: BMN 110

INTERVENTIONS:
Drug: BMN 110 — Subjects will receive a weekly 4- to 5-hour intravenous infusion of BMN 110 in 3 consecutive 12-week dosing intervals, using the following regimen:
  * Weeks 1-12: 0.1 mg/kg/week
  * Weeks 13-24: 1.0 mg/kg/week
  * Weeks 25-36: 2.0 mg/kg/week
  Subjects who complete the 36-week Dose-Escalation Period will have the option to continue drug treatment for an additional 36 to 48 weeks. Subjects continuing on treatment after the Dose-Escalation period will receive weekly 4- to 5-hour intravenous infusions of BMN 110 at a dose of 1.0 mg/kg/week.

SUMMARY:
This multicenter, open-label study is designed to assess safety, dose-response using pharmacokinetic (PK) and pharmacodynamic (PD) measures, and clinical efficacy of BMN 110 in subjects between 5 and 18 years of age, diagnosed with Mucopolysaccharidosis IVA (MPS IVA).

ELIGIBILITY:
Inclusion Criteria:

* Documented history of reduced GALNS activity relative to the normal range of the laboratory performing the assay, or documented result of molecular genetic testing confirming diagnosis of MPS IVA.
* Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 16 years, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Between 5 and 18 years of age, inclusive.
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study.
* Willing to perform all study procedures as physically possible.

Exclusion Criteria:

* Previous hematopoietic stem cell transplant (HSCT).
* Has known hypersensitivity to BMN 110 or its excipients.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Concurrent disease or condition that would interfere with study participation or safety, including, but not limited to, symptomatic cervical spine instability.
* Any condition that, in the view of the Principal Investigator (PI), places the subject at high risk of poor treatment compliance or of not completing the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Decker, MD, Study Director — BioMarin Pharmceutical Inc.
Locations (3):
- United Kingdom (3):
  - Birmingham
  - London
  - Manchester

REFERENCES:
- [Derived] Hendriksz C, Santra S, Jones SA, Geberhiwot T, Jesaitis L, Long B, Qi Y, Hawley SM, Decker C. Safety, immunogenicity, and clinical outcomes in patients with Morquio A syndrome participating in 2 sequential open-label studies of elosulfase alfa enzyme replacement therapy (MOR-002/MOR-100), representing 5 years of treatment. Mol Genet Metab. 2018 Apr;123(4):479-487. doi: 10.1016/j.ymgme.2018.02.011. Epub 2018 Feb 19. PMID 29526614
- See also: BioMarin Pharmaceutical Inc. website — http://www.bmrn.com

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN 110: Dose-Escalation Period:
  Subjects will receive a weekly 4- to 5-hour intravenous infusion of BMN 110 in 3 consecutive 12-week dosing intervals, using the following regimen:
  * Weeks 1-12: 0.1 mg/kg/week
  * Weeks 13-24: 1.0 mg/kg/week
  * Weeks 25-36: 2.0 mg/kg/week
  Continuation Period:
  Subjects who complete the 36-week Dose-Escalation Period will have the option to continue drug treatment for an additional 36 to 48 weeks. Subjects continuing on treatment after the Dose-Escalation period will receive weekly 4- to 5-hour intravenous infusions of BMN 110 at a dose of 1.0 mg/kg/week.
Period: Weeks 1-12: 0.1 mg/kg/Week
Arm/Group | BMN 110
Started | 20
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Weeks 13-24: 1.0 mg/kg/Week
Arm/Group | BMN 110
Started | 18
Completed | 18
Not Completed | 0
Period: Weeks 25-36: 2.0 mg/kg/Week
Arm/Group | BMN 110
Started | 18
Completed | 18
Not Completed | 0
Period: Continuation Period
Arm/Group | BMN 110
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- BMN 110: Dose-Escalation Period:
Arm/Group | BMN 110
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (2.89)
Age, Customized [Number; unit: participants]
  >=4 to <8 years | 10
  >=8 to <10 years | 6
  >=10 to <=18 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  Other | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in 6MWT
Description: Change from baseline in meters in 6-minute Walk Test. As a measure of endurance, a 6-minute walk test (6MWT) was performed according to the American Thoracic Society Guidelines. Patients were instructed to walk as far as possible in 6 minutes.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72
Population: Intent-to-Treat population (all subjects who enrolled in the study). Two patients were either physically (score was designated as 0 m) or developmentally (score was set to missing) unable to perform the 6MWT. The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BMN 110
Number analyzed (Participants) | 20
meters
  Week 12 Change from Baseline (n=19) | -20.7 (85.95)
  Week 24 Change from Baseline (n=17) | 16.3 (71.74)
  Week 36 Change from Baseline (n=17) | 13.8 (63.25)
  Week 48 Change from Baseline (n=17) | -4.8 (64.70)
  Week 72 Change from Baseline (n=17) | 4.0 (87.24)

2. Secondary Outcome: Change From Baseline in 3MSCT
Description: Change from baseline in the 3-minute Stair Climb Test. Patients walked up stairs that have a railing, which could be used for support, for 3 minutes, with the number of stairs climbed recorded. The test result was the number of steps climbed per minute.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72
Population: Intent-to-Treat population (all subjects who enrolled in the study). One patient was developmentally unable to perform the 3MSCT and the test scores were set to missing. The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | BMN 110
Number analyzed (Participants) | 20
steps/min
  Week 12 Change from Baseline (n=19) | 0.3 (14.07)
  Week 24 Change from Baseline (n=17) | 6.1 (8.66)
  Week 36 Change from Baseline (n=17) | 7.8 (13.69)
  Week 48 Change from Baseline (n=17) | 9.7 (14.42)
  Week 72 Change from Baseline (n=17) | 9.7 (13.91)

3. Secondary Outcome: Percent Change From Baseline in uKS
Description: Percent Change from baseline in Normalized Urine KS. The percent change was calculated (Week X value - baseline value)/baseline value *100%
Time Frame: Baseline to Weeks 12, 24, 36, 72
Population: Intent-to-Treat population (all subjects who enrolled in the study). The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: percentage of uKS
Arm/Group | BMN 110
Number analyzed (Participants) | 20
percentage of uKS
  Week 12 Percent Change from Baseline (n=19) | -23.2 (19.04)
  Week 24 Percent Change from Baseline (n=18) | -27.9 (17.92)
  Week 36 Percent Change from Baseline (n=18) | -40.6 (20.16)
  Week 72 Percent Change from Baseline (n=17) | -32.2 (17.10)

4. Secondary Outcome: Percent Change From Baseline in MVV
Description: Percent Change from baseline in Maximum Voluntary Ventilation.
Time Frame: Baseline to Weeks 12, 24, 36, 72
Population: Intent-to-Treat population (all subjects who enrolled in the study). The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: percentage of MVV
Arm/Group | BMN 110
Number analyzed (Participants) | 20
percentage of MVV
  Week 12 Percent Change from Baseline (n=14) | 9.9 (21.29)
  Week 24 Percent Change from Baseline (n=13) | 11.0 (21.48)
  Week 36 Percent Change from Baseline (n=14) | 10.5 (17.43)
  Week 72 Percent Change from Baseline (n=14) | 18.4 (20.77)

5. Secondary Outcome: Percent Change From Baseline in FVC
Description: Percent Change from baseline in Forced Vital Capacity.
Time Frame: Baseline to Weeks 12, 24, 36, 72
Population: Intent-to-Treat population (all subjects who enrolled in the study). The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: percentage of FVC
Arm/Group | BMN 110
Number analyzed (Participants) | 20
percentage of FVC
  Week 12 Percent Change from Baseline (n=18) | 3.4 (10.85)
  Week 24 Percent Change from Baseline (n=16) | 0.2 (16.60)
  Week 36 Percent Change from Baseline (n=16) | 10.7 (20.82)
  Week 72 Percent Change from Baseline (n=16) | 12.5 (14.88)

6. Primary Outcome: Subject Incidence of Treatment Emergent AEs
Description: The primary objective of the study was to evaluate the safety of weekly infusions of BMN 110 administered in escalating doses to subjects with MPS IVA.
  The safety variable incidence of TEAE is summarized.
Time Frame: Entire Study, through week 84
Measure: Number; unit: participants
Groups:
- 0.1 mg/kg/Week: Dose-Escalation Period: Weeks 1-12: 0.1 mg/kg/week
  Subjects will receive a weekly 4- to 5-hour intravenous infusion of BMN 110 0.1 mg/kg/week
- 1.0 mg/kg/Week: Dose-Escalation Period: Weeks 13-24: 1.0 mg/kg/week
  Subjects will receive a weekly 4- to 5-hour intravenous infusion of BMN 110 1.0 mg/kg/week
- 2.0 mg/kg/Week: Dose-Escalation Period: Weeks 25-36: 2.0 mg/kg/week
  Subjects will receive a weekly 4- to 5-hour intravenous infusion of BMN 110 2.0 mg/kg/week
- Continuation Period: Subjects who complete the 36-week Dose-Escalation Period will have the option to continue drug treatment for an additional 36 to 48 weeks. Subjects continuing on treatment after the Dose-Escalation period will receive weekly 4- to 5-hour intravenous infusions of BMN 110 at a dose of 1.0 mg/kg/week.
- Entire Study: Entire Study period includes both Dose-Escalation Period and Continuation Period.
Arm/Group | 0.1 mg/kg/Week | 1.0 mg/kg/Week | 2.0 mg/kg/Week | Continuation Period | Entire Study
Number analyzed (Participants) | 20 | 18 | 18 | 18 | 20
participants
  Any AEs | 18 | 18 | 17 | 17 | 20
  Any Study Drug-Related AEs | 12 | 10 | 7 | 8 | 14
  Any SAEs | 6 | 2 | 8 | 6 | 14
  Any Study Drug-Related SAEs | 2 | 1 | 2 | 1 | 4
  Any AEs During Infusion | 15 | 13 | 10 | 15 | 17
  Any SAEs During Infusion | 5 | 0 | 1 | 1 | 6
  Any AEs Causing Study Discontinuation | 1 | 0 | 0 | 0 | 1
  Any Study Drug-Related AE Causing Study Discont. | 1 | 0 | 0 | 0 | 1
  AEs Causing Permanent Study Drug Discont. | 1 | 0 | 0 | 0 | 1
  Drug-Related AE Causing Permanent StudyDrug Discon | 1 | 0 | 0 | 0 | 1
  Any SAEs Causing Study Discontinuation | 1 | 0 | 0 | 0 | 1
  Any SAEs Causing Permanent Study Drug Discont. | 1 | 0 | 0 | 0 | 1
  Study Drug-Related SAE Causing Study Discont. | 1 | 0 | 0 | 0 | 1
  StudyDrug-Related SAE Causing Permanent DrugDiscon | 1 | 0 | 0 | 0 | 1
  Death | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study Period, through 84 weeks
Description: All Adverse Events
Arm/Group | 0.1 mg/kg/Week | 1.0 mg/kg/Week | 2.0 mg/kg/Week | Continuation Period | Entire Study
Serious Adverse Events (participants affected / at risk) | 6/20 | 2/18 | 8/18 | 6/18 | 14/20
Other Adverse Events (participants affected / at risk) | 18/20 | 18/18 | 16/18 | 17/18 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.1 mg/kg/Week (N=20) | 1.0 mg/kg/Week (N=18) | 2.0 mg/kg/Week (N=18) | Continuation Period (N=18) | Entire Study (N=20)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (4)
Type I hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abscess drainage (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Catheterisation venous (Surgical and medical procedures) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Poor venous access (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.1 mg/kg/Week (N=20) | 1.0 mg/kg/Week (N=18) | 2.0 mg/kg/Week (N=18) | Continuation Period (N=18) | Entire Study (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear canal erythema (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (2) | 1 (3) | 5 (10) | 5 (16)
External ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eyelid cyst (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (3) | 1 (2) | 4 (10)
Abdominal pain upper (Gastrointestinal disorders) | 4 (8) | 1 (2) | 3 (6) | 4 (4) | 8 (20)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4) | 1 (2) | 6 (8)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 3 (5)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 4 (5)
Vomiting (Gastrointestinal disorders) | 2 (3) | 7 (7) | 4 (6) | 12 (26) | 13 (42)
Application site vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Catheter site pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Extravasation (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Implant site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4)
Implant site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Implant site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Infusion site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Pyrexia (General disorders) | 6 (6) | 9 (12) | 5 (8) | 10 (20) | 14 (46)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 5 (6)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Helminthic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lice infestation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (3) | 3 (3) | 1 (1) | 4 (6) | 8 (13)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (4)
Device migration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (2) | 1 (2) | 5 (7)
Head injury (Injury, poisoning and procedural complications) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 4 (7)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood immunoglobulin E increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Computerised tomogram (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Echocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram T wave amplitude decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nuclear magnetic resonance imaging (Investigations) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 6 (7)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Protein total abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4) | 0 (0) | 4 (4) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 4 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (3) | 1 (1) | 4 (5) | 10 (15)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 4 (8) | 2 (3) | 1 (8) | 6 (16) | 9 (35)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Balanitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7) | 3 (3) | 10 (18) | 13 (29)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 6 (6)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 4 (6)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 3 (4)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cautery to nose (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Induction of anaesthesia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (4)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Poor venous access (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish any data prior to multi-centre publication. If publication related to sub-sets of data shall make reference to the relevant multi-centre publication. PI agrees to submit data to Sponsor for review and comment 60 days prior to publication. During review period, Sponsor may request that publication be delayed for up to 6 months from date of first submission to Sponsor in order for Sponsor to take steps to protect its proprietary information.